CLINICAL TRIAL: NCT03967054
Title: Repeat Ivermectin Mass Drug Administrations for MALaria Control II (RIMDAMAL II): a Double-blind, Cluster-randomized Control Trial for Integrated Control of Malaria
Brief Title: Repeat Ivermectin Mass Drug Administrations for MALaria Control II
Acronym: RIMDAMAL II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brian Foy (Other)
Collaborators: Yale University (Other); Institut de Recherche en Sciences de la Sante-Direction Regionale de l'Ouest (Other Government); Radboud University Medical Center (Other); PATH (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Brian Foy, Professor, Colorado State University
Organization: Colorado State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1691; U01AI138910 (NIH)
Record Dates: First submitted 2019-05-24; First posted 2019-05-30 (Actual); Results first posted 2024-01-11 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Malaria
Keywords: mosquito; ivermectin; Anopheles; Plasmodium
MeSH Terms: conditions — Malaria | interventions — Ivermectin

STUDY DESIGN:
Intervention Model Description: Parallel-assignment trial with two arms randomized in a 1:1 ratio.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study pharmacist in charge of the drug stock room will originate the masking and maintain the masking from all other investigators. The masking codes will be written on three paper copies and put in identical and sealed opaque envelopes, which will be kept in three different areas.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ivermectin mass drug administration (Experimental): Ivermectin given monthly from July-October (4 times) as a 3-day course of 300 µg/kg/day to all eligible persons per exclusion/inclusion criteria. Per package insert, dosing of IVM will be according to height to approximate weight: 90-119 cm = 1 tablet/day for 3 days; 120-140 cm = 2 tablets/day for 3 days; 141-158 cm = 3 tablets/day for 3 days; >158 cm = 4 tablet/day for 3 days.
  Interventions: Drug: Ivermectin
- Placebo mass administration (Placebo Comparator): Placebo given monthly from July-October (4 times) as a 3-day course to all eligible persons per exclusion/inclusion criteria. Dosing of placebo will be according to height to approximate weight: 90-119 cm = 1 tablet/day for 3 days; 120-140 cm = 2 tablets/day for 3 days; 141-158 cm = 3 tablets/day for 3 days; >158 cm = 4 tablet/day for 3 days.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Ivermectin — Ivermectin (6 mg tablet) given monthly from July-October each rainy season as a 3-day course of approximately 300 mcg/kg/day as estimated by height bands.
  Other Names: Iver P
  Arms: Ivermectin mass drug administration
Drug: Placebo oral tablet — placebo in the same size, color and shape at the ivermectin tablet
  Arms: Placebo mass administration

SUMMARY:
RIMDAMAL II is a double-blind, cluster randomized trial in Burkina Faso designed to test whether repeated ivermectin mass drug administrations, integrated into a monthly delivery platform with standard malaria control measures of seasonal malaria chemoprevention and insecticide-treated bed net distribution in the Sahel, will reduce childhood malaria incidence.

DETAILED DESCRIPTION:
The RIMDAMAL II trial is designed to determine the efficacy of adding seasonal ivermectin mass drug administrations to the standard-policy malaria control measures in the Sahel (seasonal malaria chemoprevention in children, maximum long-lasting insecticidal net coverage, intermittent preventive treatment in pregnancy), for reducing the incidence of uncomplicated malaria episodes in enrolled village children (≤ 10 years of age) assessed by active case surveillance. The investigators will also examine the safety of the intervention, as well as entomological and parasitological endpoints. This is a double-blind, cluster randomized trial in that will occur in villages in southwestern Burkina Faso over two consecutive rainy seasons. For the intervention, mass administration of ivermectin or placebo will be given monthly over 4 months of each rainy season to the eligible village population, each as 3-day course of 300 µg/kg/day. These mass drug administrations will occur simultaneously with the distribution of seasonal malaria chemoprevention drugs on the same monthly schedule to eligible children aged 3-59 months.

ELIGIBILITY:
Inclusion Criteria (for being enrolled in the study):

* Residence in selected study village
* Able to understand the information and willing to give consent or assent (age 12-18) and parent/guardian consent if study participant age is < 18 years of age.

Exclusion Criteria (for participating in the intervention [ivermectin or placebo MDA]):

* Residence outside of the study village
* Height < 90 cm (*note: if subject becomes ≥90cm over course the trial, this exclusion criteria will no longer be valid in subsequent MDA)
* Current treatment with SP+AQ as part of SMC (restricted to children 3-59 months old) (*note: if subject discontinuous SP+AQ treatment because they become older than 59 months over course the trial, this exclusion criteria will no longer be valid in subsequent MDA)
* Permanent disability or serious medical illness that prevents or impedes study participation and/or comprehension
* Pregnancy (screened for in women of child-bearing age [ages 15-45] using a pregnancy urine rapid test [e.g. SD Bioline hCG] the week prior to each MDA)
* Breast feeding if infant is within 1 week of birth
* Known allergy to ivermectin
* Possibility of Loa loa infection as assessed by travel history to Angola, Cameroon, Chad, Central African Republic, Congo, Democratic Republic of Congo, Equatorial Guinea, Ethiopia, Gabon, Nigeria, and Sudan.
* Enrolled in any other active clinical trials

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4124 (Actual)
Dates: Start 2019-07-13 (Actual); Primary Completion 2020-11-08 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian D. Foy, PhD, Principal Investigator — Colorado State University; Sunil Parikh, MD, Principal Investigator — Yale University
Locations (1):
- Institut de Recherche en Sciences de la Sante, Diébougou, Sud-Ouest Region, Burkina Faso

IPD SHARING:
Plan to Share IPD: Yes
Data collected from this study, including de-identified individual participant data, will be made available upon publication to members of the scientific and medical community for non-commercial use only, upon email request to the corresponding author. The finalized study protocol, statistical analysis plan, and informed consent forms will be made available on ClinicalTrials.gov.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 6 mos of publication of the primary outcomes of the study.

REFERENCES:
- [Derived] Some AF, Some A, Sougue E, Ouedraogo COW, Da O, Dah SR, Nikiema F, Magalhaes T, Gray LI, Finical W, Pugh G, Lado P, Randall JC, Burton TA, Ring ME, Leon AS, Colt M, Li F, Wang K, Wade M, Lier AJ, Richards K, Sproch H, Zhang E, Ellman J, Achebe I, Jackson CL, Xiao M, Wu EJ, Bousema T, Slater HC, Foy BD, Parikh S, Dabire RK. Safety and efficacy of repeat ivermectin mass drug administrations for malaria control (RIMDAMAL II): a phase 3, double-blind, placebo-controlled, cluster-randomised, parallel-group trial. Lancet Infect Dis. 2025 Jul;25(7):737-750. doi: 10.1016/S1473-3099(24)00751-5. Epub 2025 Feb 4. PMID 39919778
- [Derived] Foy BD, Some A, Magalhaes T, Gray L, Rao S, Sougue E, Jackson CL, Kittelson J, Slater HC, Bousema T, Da O, Coulidiaty AGV, Colt M, Wade M, Richards K, Some AF, Dabire RK, Parikh S. Repeat Ivermectin Mass Drug Administrations for Malaria Control II: Protocol for a Double-blind, Cluster-Randomized, Placebo-Controlled Trial for the Integrated Control of Malaria. JMIR Res Protoc. 2023 Mar 20;12:e41197. doi: 10.2196/41197. PMID 36939832

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential clusters (villages) within the Diebougou Health district, Burkina Faso, were identified from a catchment area based on access, safety of the study team, potential for contamination, and cluster size, and invited to participant via an extensive community engagement process.
Units Other Than Participants: villages
Period: Overall Study
Arm/Group | Ivermectin Mass Drug Administration | Placebo Mass Administration
Started | 2191; 7 villages | 1933; 7 villages
Completed | 2191; 7 villages | 1933; 7 villages
Not Completed | 0; 0 villages | 0; 0 villages

BASELINE CHARACTERISTICS:
Population: All participants were evaluated for adverse events, but only eligible participants participated in the intervention (ivermectin or placebo mass administration. The primary outcome measure comes only from malaria incidence measurements within a cohort of village children <= 10 years of age (1531 participants).
Groups:
- Total: Total of all reporting groups
Arm/Group | Ivermectin Mass Drug Administration | Placebo Mass Administration | Total
Number analyzed (Participants) | 2191 | 1933 | 4124
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 17 [7 to 36] | 15 [6 to 35] | 16 [7 to 36]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1100 | 1024 | 2124
  Male | 1091 | 909 | 2000
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2191 | 1933 | 4124
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Residents of villages located in the Diebougou health district in southwestern Burkina Faso
  participants
    Burkina Faso | 2191 | 1933 | 4124

OUTCOME MEASURES:

1. Primary Outcome: Malaria Incidence
Description: Incidence of malaria episodes in enrolled village children ≤ 10 years of age
Time Frame: up to 8 months
Population: The primary outcome measure comes only from malaria incidence measurements within a cohort of village children (1531). It is not a measure of malaria incidence from all enrolled participants from the study villages. The majority of participants (1133/1531) within the child cohort were evaluated in both years, meaning that they contributed a malaria case count for both year 1 and year 2.
Measure: Mean (95% Confidence Interval); unit: Malaria cases per person-week
Arm/Group | Ivermectin Mass Drug Administration | Placebo Mass Administration
Number analyzed (Participants) | 795 | 736
Malaria cases per person-week | 0.0176 [0.0124 to 0.0252] | 0.0183 [0.0128 to 0.0262]

2. Secondary Outcome: Adverse Events
Description: Number adverse events among the study population over the course of the intervention period. Note, this number includes all malaria cases that were part of the primary outcome that occurred in the cohort of children that were actively assessed for malaria on a weekly basis during the intervention.
Time Frame: up to 8 months
Measure: Number; unit: adverse events
Arm/Group | Ivermectin Mass Drug Administration | Placebo Mass Administration
Number analyzed (Participants) | 2191 | 1933
adverse events | 438 | 402

3. Secondary Outcome: Survival Rate of Blood Fed Mosquitoes
Description: Number of Blood Fed Mosquitoes Alive For 3 Days After Capture
Time Frame: up to 8 months
Population: This analysis population is not human participants but mosquitoes captured from participants' homes. These are blood fed Anopheles gambiae s.l. mosquitoes captured indoors in participants' home 1 week following each mass drug administration.
Measure: Count of Units; unit: mosquitoes
Units Other Than Participants: mosquitoes
Arm/Group | Ivermectin Mass Drug Administration | Placebo Mass Administration
Number analyzed (Participants) | 2191 | 1933
Number analyzed (mosquitoes) | 660 | 1258
mosquitoes | 399 | 896

ADVERSE EVENTS:
Time Frame: Adverse events were recorded over the intervention period, which occurred over two 4-month intervals of 2 consecutive rainy seasons in 2019 and 2020 (8 total months).
Arm/Group | Ivermectin Mass Drug Administration | Placebo Mass Administration
All-Cause Mortality (participants affected / at risk) | 6/2191 | 3/1933
Serious Adverse Events (participants affected / at risk) | 8/2191 | 6/1933
Other Adverse Events (participants affected / at risk) | 430/2191 | 396/1933
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ivermectin Mass Drug Administration (N=2191) | Placebo Mass Administration (N=1933)
cellulitis (Infections and infestations) | 1 (1) | 1 (1)
nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1)
spontaneous abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
liver cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
liver failure (Hepatobiliary disorders) | 1 (1) | 1 (1)
head trauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
sepsis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ivermectin Mass Drug Administration (N=2191) | Placebo Mass Administration (N=1933)
malaria (Infections and infestations) | 355 (466) | 308 (436)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
abcess (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (6)
bite wound (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
blurry vision (Eye disorders) | 1 (1) | 0 (0)
breast tenderness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
breast cancer (Reproductive system and breast disorders) | 1 (1) | 0 (0)
burn (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
cellulitis (Infections and infestations) | 0 (0) | 1 (1)
chills (General disorders) | 0 (0) | 1 (1)
conjunctivitis (Eye disorders) | 1 (1) | 2 (2)
cough (Infections and infestations) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 6 (6) | 7 (7)
dizziness (Ear and labyrinth disorders) | 5 (5) | 0 (0)
dysphagia (Gastrointestinal disorders) | 1 (1) | 2 (2)
edema (General disorders) | 2 (2) | 1 (1)
failure to thrive (General disorders) | 1 (1) | 0 (0)
fatigue (General disorders) | 2 (2) | 0 (0)
fever (General disorders) | 11 (11) | 10 (10)
gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
gastroenteritis (Gastrointestinal disorders) | 3 (3) | 1 (1)
gastrointestinal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 6 (6) | 6 (6)
hives (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
hypersensitivity (General disorders) | 1 (1) | 0 (0)
injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
lower back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
myalgia (General disorders) | 1 (1) | 2 (2)
otalgia (Ear and labyrinth disorders) | 0 (0) | 6 (6)
otitis media (Ear and labyrinth disorders) | 1 (1) | 3 (3)
pain (General disorders) | 0 (0) | 5 (5)
pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
procedural (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
pruritis (Skin and subcutaneous tissue disorders) | 9 (9) | 20 (20)
rash (Skin and subcutaneous tissue disorders) | 5 (5) | 12 (12)
snake bite (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
trauma (Injury, poisoning and procedural complications) | 4 (4) | 7 (7)
upper respiratory infection (Infections and infestations) | 13 (13) | 26 (29)
vertigo (Ear and labyrinth disorders) | 3 (3) | 0 (0)
vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-02-29): https://cdn.clinicaltrials.gov/large-docs/54/NCT03967054/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT03967054/SAP_001.pdf